CLINICAL TRIAL: NCT05557929
Title: Cardiopulmonary Exercise Testing Parameters' Variability During Long and Short Interdialytic Intervals in Hemodialysis Patients.
Brief Title: Cardiopulmonary Exercise Testing Parameters' Variability in Hemodialysis Patients.
Status: Completed | Type: Observational
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Other Study IDs: ΔΔ4878
Record Dates: First submitted 2022-09-20; First posted 2022-09-28 (Actual); Last update posted 2023-08-22 (Actual); Status verified 2023-08

CONDITIONS: Chronic Kidney Disease Requiring Chronic Dialysis; Chronic Kidney Diseases
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Other | Time Perspective: Other
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Hemodialysis patients: The present study will comparatively evaluate a series of parameters (measured with cardiopulmonary exercise testing, spirometry, heart ultrasound, lung ultrasound and bioelectrical impedance analysis) in end-stage kidney disease patients undergoing hemodialysis between the end of the long and the end of the short interdialytic interval. The primary aim of the study is the evaluation of cardiorespiratory fitness - cardiovascular reserve assessed with cardiopulmonary exercise testing at these time points.
- Controls without CKD: Controls without CKD will be evaluated with cardiopulmonary exercise testing, spirometry, heart ultrasound, lung ultrasound and bioelectrical impedance analysis at one time point (baseline visit)

SUMMARY:
Chronic kidney disease (CKD), especially end-stage kidney disease (ESKD), is associated with increased risk for cardiovascular events and all-cause mortality. Exercise intolerance as well as reduced cardiovascular reserve are extremely common in patients with CKD. Cardiopulmonary exercise testing (CPET) is a non-invasive, dynamic technique that provides an integrative evaluation of cardiovascular, pulmonary, neuropsychological and metabolic function during maximal or submaximal exercise, allowing the evaluation of functional reserves of these systems. CPET is currently considered to be the gold-standard for identifying exercise limitation and differentiating its causes. It has been widely used in several medical fields for risk stratification, clinical evaluation and other applications. However, the use of CPET in assessment of exercise intolerance in everyday nephrology practice is limited. Hence, this is the first study possible differences in CPET's parameters during long and short interdialytic intervals in hemodialysis patients.

DETAILED DESCRIPTION:
This is an observational study with a cross-over design performed in the Department of Nephrology and the Third Department of Cardiology in Hippokration Hospital of Thessaloniki in Greece. For the purposes of this study, hemodialysis patients fulfilling the inclusion/exclusion criteria, as well as controls without CKD, were invited to participate. All included patients signed a written informed consent form. The study protocol was approved by the Ethics Committee of the School of Medicine, Aristotle University of Thessaloniki. All procedures and evaluations are performed according to the Declaration of Helsinki 2013 Amendment.

Baseline evaluation includes the recording of demographics and anthropometric characteristics, medical history, concomitant medications and dialysis-related parameters, as well as physical examination and venous blood sampling for routine laboratory tests. Hemodialysis patients will be evaluated at two time points (at the end of the long and at the end of the short interdialytic interval), while controls at one time point. All the participants will undergo spirometry, CPET, cardiac ultrasound, lung ultrasound and bioelectrical impedance analysis.

ELIGIBILITY:
Inclusion Criteria:

* Hemodialysis patients aged >18 years.
* Patients with a total duration of hemodialysis >3 months.
* Patients enrolled in a dialysis program that includes three sessions per week.
* Hemodialysis patients who are capable of exercising on a cycle ergometer.
* Hemodialysis patients who are capable of understanding and providing written, signed consent to participate in the study

Exclusion Criteria:

Absolute and relative contraindications for performing CPET according to the American Thoracic Society (ATS) and the American College of Chest Physicians (ACCP), such as

* Acute myocardial infarction (3-5 days)
* Unstable angina
* Uncontrolled arrhythmias causing symptoms or haemodynamic compromise
* Syncope
* Active endocarditis
* Acute myocarditis or pericarditis
* Symptomatic severe aortic stenosis
* Uncontrolled heart failure
* Acute pulmonary embolus or pulmonary infarction
* Thrombosis of lower extremities
* Suspected dissecting aneurysm
* Uncontrolled asthma
* Pulmonary oedema
* Acute non-cardiopulmonary disorder that may affect exercise performance or be aggravated by exercise (ie, infection, renal failure, thyrotoxicosis)
* Mental impairment leading to inability to cooperate
* Orthopaedic impairment that compromises exercise performance
* Electrolyte abnormalities
* Advanced or complicated pregnancy...

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Hemodialysis patients evaluated during the long and the shord dialysis interval Controls without kidney failure
Sampling Method: Non-Probability Sample
Enrollment: 28 (Actual)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-07-28 (Actual); Study Completion 2023-07-28 (Actual)

PRIMARY OUTCOMES:
Difference in VO2peak (ml/min/kg) | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in VO2peak (ml/min/kg) assessed with CPET between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in VO2peak ((ml/min) | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in VO2peak (ml/min) assessed with CPET between long and short Interdialytic Interval in Hemodialysis Patients.

SECONDARY OUTCOMES:
Difference in Maximum workload (Watt) | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in Maximum workload (Watt) assessed with CPET between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in VCO2 (ml/min) | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in VCO2 (ml/min) assessed with CPET between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in Heart Rate (bpm) | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in Heart Rate (bpm) assessed with CPET between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in O2 pulse | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in O2 pulse assessed with CPET between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in VE (L/min) | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in VE (L/min) assessed with CPET between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in Tidal Volume, VT (ml) | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in Tidal Volume, VT (ml) assessed with CPET between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in Respiratory Rate, RR | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in Respiratory Rate, RR assessed with CPET between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in PETCO2 (mmHg) | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in PETCO2 (mmHg) assessed with CPET between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in PETO2 (mmHg) | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in PETO2 (mmHg) assessed with CPET between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in VE/VCO2 | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in VE/VCO2 assessed with CPET between long and short Interdialytic Interval in Hemodialysis Patients.

OTHER OUTCOMES:
Difference in Forced expiratory volume in one second, FEV1 | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in Forced expiratory volume in one second, FEV1 assessed with Spirometry between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in Forced vital capacity, FVC | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in Forced vital capacity, FVC assessed with Spirometry between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in FEV1/FVC | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in FEV1/FVC assessed with Spirometry between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in Total lung capacity, TLC | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in Total lung capacity, TLC assessed with Spirometry between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in Residual volume, RV | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in Residual volume, RV assessed with Spirometry between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in Left ventricular mass index, LVMI | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in Left ventricular mass index, LVMI assessed with Heart Ultrasound between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in Left ventricular end-systolic volume, LVESV | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in Left ventricular end-systolic volume, LVESV assessed with Heart Ultrasound between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in Left ventricular end-diastolic volume, LVEDV | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in Left ventricular end-diastolic volume, LVEDV assessed with Heart Ultrasound between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in Global longitudinal strain, GLS | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in Global longitudinal strain, GLS assessed with Heart Ultrasound between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in Right ventricular free wall - RVFW GLS | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in Right ventricular free wall - RVFW GLS assessed with Heart Ultrasound between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in Tricuspid annular plane systolic excursion - TAPSE | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in Tricuspid annular plane systolic excursion - TAPSE assessed with Heart Ultrasound between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in Tissue Doppler imaging - TDI S | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in Tissue Doppler imaging - TDI S assessed with Heart Ultrasound between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in Pulmonary artery systolic pressure - PASP | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in Pulmonary artery systolic pressure - PASP assessed with Heart Ultrasound between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in E/e | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in E/e assessed with Heart Ultrasound between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in E/A | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in E/A assessed with Heart Ultrasound between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in Left atrial volume index - LAVi | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in Left atrial volume index - LAVi assessed with Heart Ultrasound between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in Left ventricular ejection fraction, LVEF | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in Left ventricular ejection fraction, LVEF assessed with Heart Ultrasound between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in Diameter of the inferior vena cava, IVC | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in Diameter of the inferior vena cava, IVC assessed with Heart Ultrasound between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in B- lines' number | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in B- lines' number assessed with Lung Ultrasound between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in Total body water, TBW | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in Total body water, TBW assessed with Bioelectrical impedance analysis between long and short Interdialytic Interval in Hemodialysis Patients.
Difference in Fat-free mass, FFM | Two-week time frame between the study evaluation time points (before dialysis session after the long interdialytic interval versus before dialysis session after the short interdialytic interval)
  Difference in Fat-free mass, FFM assessed with Bioelectrical impedance analysis between long and short Interdialytic Interval in Hemodialysis Patients.

CONTACTS AND LOCATIONS:
Overall Officials: Pantelis Sarafidis, Professor, Principal Investigator — Aristotle University of Thessaloniki, Greece
Locations (1):
- Hippokration General Hospital of Thessaloniki, Aristotle University of Thessaloniki, Thessaloniki, Thessalonikis, Greece

REFERENCES:
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- [Background] Andrassy KM. Comments on 'KDIGO 2012 Clinical Practice Guideline for the Evaluation and Management of Chronic Kidney Disease'. Kidney Int. 2013 Sep;84(3):622-3. doi: 10.1038/ki.2013.243. No abstract available. PMID 23989362
- [Background] Foley RN, Parfrey PS, Sarnak MJ. Clinical epidemiology of cardiovascular disease in chronic renal disease. Am J Kidney Dis. 1998 Nov;32(5 Suppl 3):S112-9. doi: 10.1053/ajkd.1998.v32.pm9820470. No abstract available.
- [Background] London GM, Drueke TB. Atherosclerosis and arteriosclerosis in chronic renal failure. Kidney Int. 1997 Jun;51(6):1678-95. doi: 10.1038/ki.1997.233. No abstract available. PMID 9186855
- [Background] Wolf M. Forging forward with 10 burning questions on FGF23 in kidney disease. J Am Soc Nephrol. 2010 Sep;21(9):1427-35. doi: 10.1681/ASN.2009121293. Epub 2010 May 27. PMID 20507943
- [Background] Bernheim J, Benchetrit S. The potential roles of FGF23 and Klotho in the prognosis of renal and cardiovascular diseases. Nephrol Dial Transplant. 2011 Aug;26(8):2433-8. doi: 10.1093/ndt/gfr208. Epub 2011 May 4. PMID 21543658
- [Background] Go AS, Chertow GM, Fan D, McCulloch CE, Hsu CY. Chronic kidney disease and the risks of death, cardiovascular events, and hospitalization. N Engl J Med. 2004 Sep 23;351(13):1296-305. doi: 10.1056/NEJMoa041031. PMID 15385656
- [Background] de Jager DJ, Grootendorst DC, Jager KJ, van Dijk PC, Tomas LM, Ansell D, Collart F, Finne P, Heaf JG, De Meester J, Wetzels JF, Rosendaal FR, Dekker FW. Cardiovascular and noncardiovascular mortality among patients starting dialysis. JAMA. 2009 Oct 28;302(16):1782-9. doi: 10.1001/jama.2009.1488. PMID 19861670
- [Background] Georgianos PI, Sarafidis PA. Pro: Should we move to more frequent haemodialysis schedules? Nephrol Dial Transplant. 2015 Jan;30(1):18-22. doi: 10.1093/ndt/gfu381. Epub 2014 Dec 23. PMID 25538158
- [Background] Saran R, Li Y, Robinson B, Abbott KC, Agodoa LY, Ayanian J, Bragg-Gresham J, Balkrishnan R, Chen JL, Cope E, Eggers PW, Gillen D, Gipson D, Hailpern SM, Hall YN, He K, Herman W, Heung M, Hirth RA, Hutton D, Jacobsen SJ, Kalantar-Zadeh K, Kovesdy CP, Lu Y, Molnar MZ, Morgenstern H, Nallamothu B, Nguyen DV, O'Hare AM, Plattner B, Pisoni R, Port FK, Rao P, Rhee CM, Sakhuja A, Schaubel DE, Selewski DT, Shahinian V, Sim JJ, Song P, Streja E, Kurella Tamura M, Tentori F, White S, Woodside K, Hirth RA. US Renal Data System 2015 Annual Data Report: Epidemiology of Kidney Disease in the United States. Am J Kidney Dis. 2016 Mar;67(3 Suppl 1):Svii, S1-305. doi: 10.1053/j.ajkd.2015.12.014. No abstract available. PMID 26925525
- [Background] Bleyer AJ, Russell GB, Satko SG. Sudden and cardiac death rates in hemodialysis patients. Kidney Int. 1999 Apr;55(4):1553-9. doi: 10.1046/j.1523-1755.1999.00391.x. PMID 10201022
- [Background] Foley RN, Gilbertson DT, Murray T, Collins AJ. Long interdialytic interval and mortality among patients receiving hemodialysis. N Engl J Med. 2011 Sep 22;365(12):1099-107. doi: 10.1056/NEJMoa1103313. PMID 21992122
- [Background] Zhang H, Schaubel DE, Kalbfleisch JD, Bragg-Gresham JL, Robinson BM, Pisoni RL, Canaud B, Jadoul M, Akiba T, Saito A, Port FK, Saran R. Dialysis outcomes and analysis of practice patterns suggests the dialysis schedule affects day-of-week mortality. Kidney Int. 2012 Jun;81(11):1108-15. doi: 10.1038/ki.2011.481. Epub 2012 Feb 1. PMID 22297673
- [Background] Tsilonis K, Sarafidis PA, Kamperidis V, Loutradis C, Georgianos PI, Imprialos K, Ziakas A, Sianos G, Nikolaidis P, Lasaridis AN, Karvounis H. Echocardiographic Parameters During Long and Short Interdialytic Intervals in Hemodialysis Patients. Am J Kidney Dis. 2016 Nov;68(5):772-781. doi: 10.1053/j.ajkd.2016.06.017. Epub 2016 Aug 18. PMID 27545351
- [Background] Koutroumbas G, Georgianos PI, Sarafidis PA, Protogerou A, Karpetas A, Vakianis P, Raptis V, Liakopoulos V, Panagoutsos S, Syrganis C, Passadakis P. Ambulatory aortic blood pressure, wave reflections and pulse wave velocity are elevated during the third in comparison to the second interdialytic day of the long interval in chronic haemodialysis patients. Nephrol Dial Transplant. 2015 Dec;30(12):2046-53. doi: 10.1093/ndt/gfv090. Epub 2015 Apr 28. PMID 25920919
- [Background] Pun PH. The interplay between CKD, sudden cardiac death, and ventricular arrhythmias. Adv Chronic Kidney Dis. 2014 Nov;21(6):480-8. doi: 10.1053/j.ackd.2014.06.007. Epub 2014 Oct 24. PMID 25443573
- [Background] Sarafidis PA, Bakris GL. Cardiovascular disease in CKD in 2014: new insights into cardiovascular risk factors and outcomes. Nat Rev Nephrol. 2015 Feb;11(2):70-2. doi: 10.1038/nrneph.2014.242. Epub 2014 Dec 16. PMID 25511758
- [Background] Da J, Xie X, Wolf M, Disthabanchong S, Wang J, Zha Y, Lv J, Zhang L, Wang H. Serum Phosphorus and Progression of CKD and Mortality: A Meta-analysis of Cohort Studies. Am J Kidney Dis. 2015 Aug;66(2):258-65. doi: 10.1053/j.ajkd.2015.01.009. Epub 2015 Mar 21. PMID 25804679
- [Background] Georgianos PI, Sarafidis PA, Sinha AD, Agarwal R. Adverse effects of conventional thrice-weekly hemodialysis: is it time to avoid 3-day interdialytic intervals? Am J Nephrol. 2015;41(4-5):400-8. doi: 10.1159/000435842. Epub 2015 Jun 27. PMID 26139107
- [Background] Cerasola G, Nardi E, Palermo A, Mule G, Cottone S. Epidemiology and pathophysiology of left ventricular abnormalities in chronic kidney disease: a review. J Nephrol. 2011 Jan-Feb;24(1):1-10. doi: 10.5301/jn.2010.2030. PMID 20437402
- [Background] Segall L, Nistor I, Covic A. Heart failure in patients with chronic kidney disease: a systematic integrative review. Biomed Res Int. 2014;2014:937398. doi: 10.1155/2014/937398. Epub 2014 May 15. PMID 24959595
- [Background] Johansen KL, Kaysen GA, Dalrymple LS, Grimes BA, Glidden DV, Anand S, Chertow GM. Association of physical activity with survival among ambulatory patients on dialysis: the Comprehensive Dialysis Study. Clin J Am Soc Nephrol. 2013 Feb;8(2):248-53. doi: 10.2215/CJN.08560812. Epub 2012 Nov 2. PMID 23124787
- [Background] Sietsema KE, Amato A, Adler SG, Brass EP. Exercise capacity as a predictor of survival among ambulatory patients with end-stage renal disease. Kidney Int. 2004 Feb;65(2):719-24. doi: 10.1111/j.1523-1755.2004.00411.x. PMID 14717947
- [Background] Ting SM, Iqbal H, Kanji H, Hamborg T, Aldridge N, Krishnan N, Imray CH, Banerjee P, Bland R, Higgins R, Zehnder D. Functional cardiovascular reserve predicts survival pre-kidney and post-kidney transplantation. J Am Soc Nephrol. 2014 Jan;25(1):187-95. doi: 10.1681/ASN.2013040348. Epub 2013 Nov 14. PMID 24231666
- [Background] Heiwe S, Clyne N, Dahlgren MA. Living with chronic renal failure: patients' experiences of their physical and functional capacity. Physiother Res Int. 2003;8(4):167-77. doi: 10.1002/pri.287. PMID 14730721
- [Background] Heiwe S, Jacobson SH. Exercise training for adults with chronic kidney disease. Cochrane Database Syst Rev. 2011 Oct 5;2011(10):CD003236. doi: 10.1002/14651858.CD003236.pub2. PMID 21975737
- [Background] Albouaini K, Egred M, Alahmar A, Wright DJ. Cardiopulmonary exercise testing and its application. Postgrad Med J. 2007 Nov;83(985):675-82. doi: 10.1136/hrt.2007.121558. PMID 17989266
- [Background] Boutou AK, Pitsiou GG, Argyropoulou P. Non-invasive markers of pulmonary hypertension in interstitial lung disease: is cardiopulmonary exercise testing the Holy Grail? Respirology. 2014 Jul;19(5):621-2. doi: 10.1111/resp.12321. Epub 2014 May 15. No abstract available. PMID 24831928
- [Background] Stavrou V, Bardaka F, Karetsi E, Daniil Z, Gourgoulianis KI. Brief Review: Ergospirometry in Patients with Obstructive Sleep Apnea Syndrome. J Clin Med. 2018 Jul 31;7(8):191. doi: 10.3390/jcm7080191. PMID 30065219
- [Background] ERS Task Force; Palange P, Ward SA, Carlsen KH, Casaburi R, Gallagher CG, Gosselink R, O'Donnell DE, Puente-Maestu L, Schols AM, Singh S, Whipp BJ. Recommendations on the use of exercise testing in clinical practice. Eur Respir J. 2007 Jan;29(1):185-209. doi: 10.1183/09031936.00046906. PMID 17197484
- [Background] Ferrazza AM, Martolini D, Valli G, Palange P. Cardiopulmonary exercise testing in the functional and prognostic evaluation of patients with pulmonary diseases. Respiration. 2009;77(1):3-17. doi: 10.1159/000186694. Epub 2009 Jan 14. PMID 19145106
- [Background] Carlisle J, Swart M. Mid-term survival after abdominal aortic aneurysm surgery predicted by cardiopulmonary exercise testing. Br J Surg. 2007 Aug;94(8):966-9. doi: 10.1002/bjs.5734. PMID 17440956
- [Background] Gitt AK, Wasserman K, Kilkowski C, Kleemann T, Kilkowski A, Bangert M, Schneider S, Schwarz A, Senges J. Exercise anaerobic threshold and ventilatory efficiency identify heart failure patients for high risk of early death. Circulation. 2002 Dec 10;106(24):3079-84. doi: 10.1161/01.cir.0000041428.99427.06. PMID 12473555
- [Background] Older P, Hall A, Hader R. Cardiopulmonary exercise testing as a screening test for perioperative management of major surgery in the elderly. Chest. 1999 Aug;116(2):355-62. doi: 10.1378/chest.116.2.355. PMID 10453862
- [Background] Older P, Smith R, Courtney P, Hone R. Preoperative evaluation of cardiac failure and ischemia in elderly patients by cardiopulmonary exercise testing. Chest. 1993 Sep;104(3):701-4. doi: 10.1378/chest.104.3.701. PMID 8365279
- [Background] Wasserman K, Hansen JE, Sue DY, et al. Principles of exercise testing and interpretation: including pathophysiology and clinical applications. Philadelphia (PA): Lipincott, Williams and Wilkins; 2005.
- [Background] American Thoracic Society; American College of Chest Physicians. ATS/ACCP Statement on cardiopulmonary exercise testing. Am J Respir Crit Care Med. 2003 Jan 15;167(2):211-77. doi: 10.1164/rccm.167.2.211. No abstract available. PMID 12524257
- [Background] Ting SM, Hamborg T, McGregor G, Oxborough D, Lim K, Koganti S, Aldridge N, Imray C, Bland R, Fletcher S, Krishnan NS, Higgins RM, Townend J, Banerjee P, Zehnder D. Reduced Cardiovascular Reserve in Chronic Kidney Failure: A Matched Cohort Study. Am J Kidney Dis. 2015 Aug;66(2):274-84. doi: 10.1053/j.ajkd.2015.02.335. Epub 2015 Apr 18. PMID 25900597
- [Background] Rogan A, McCarthy K, McGregor G, Hamborg T, Evans G, Hewins S, Aldridge N, Fletcher S, Krishnan N, Higgins R, Zehnder D, Ting SM. Quality of life measures predict cardiovascular health and physical performance in chronic renal failure patients. PLoS One. 2017 Sep 14;12(9):e0183926. doi: 10.1371/journal.pone.0183926. eCollection 2017. PMID 28910330
- [Background] Habedank D, Schefold JC, Bernhardt C, Karhausen T, Doehner W, Anker SD, Reinke P. Vasodilation and Exercise Capacity in Patients with End-Stage Renal Disease: A Prospective Proof-of-Concept Study. Cardiorenal Med. 2016 Nov;7(1):50-59. doi: 10.1159/000449174. Epub 2016 Sep 21. PMID 27994602
- [Background] Angell J, Dodds N, Darweish-Mednuik AM, Lewis S, Pyke M, Mitchell DC, Hamilton K, White P, Tolchard S. Characterising recovery from renal transplantation and live-related donation using cardiopulmonary exercise testing. Disabil Rehabil. 2021 Jun;43(12):1692-1698. doi: 10.1080/09638288.2019.1674387. Epub 2019 Oct 10. PMID 31600094
- [Background] Lim K, Ting SMS, Hamborg T, McGregor G, Oxborough D, Tomkins C, Xu D, Thadhani R, Lewis G, Bland R, Banerjee P, Fletcher S, Krishnan NS, Higgins R, Zehnder D, Hiemstra TF. Cardiovascular Functional Reserve Before and After Kidney Transplant. JAMA Cardiol. 2020 Apr 1;5(4):420-429. doi: 10.1001/jamacardio.2019.5738. PMID 32022839
- [Derived] Pella E, Boulmpou A, Boutou A, Theodorakopoulou MP, Haddad N, Karpetas A, Giamalis P, Papagianni A, Papadopoulos CE, Vassilikos V, Sarafidis P. Different Interdialytic Intervals and Cardiorespiratory Fitness in Patients Undergoing Hemodialysis. Clin J Am Soc Nephrol. 2024 Jun 1;19(6):732-742. doi: 10.2215/CJN.0000000000000435. Epub 2024 Feb 26. PMID 38407848